CLINICAL TRIAL: NCT07288905
Title: The Feasibility and Effects of Exercise Training Combined With Blood Flow Restriction Training on Exercise Capacity and Exercise Tolerance in Patients With Chronic Kidney Disease
Brief Title: Exploring the Effects of Exercise Combined With BFRT on Healthy and Patients With CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kun-Ling Tsai, Professor and Chair, Department of Physical Therapy, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-ER-113-450
Record Dates: First submitted 2025-11-16; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise; Blood Flow Restriction Therapy; Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- healthy (Experimental): We will provide BFR combined with exercise
  Interventions: Behavioral: Aerobic exercise; Behavioral: Blood flow restriction; Behavioral: Resistance exercise; Behavioral: Disease and exercise suggestion
- CKD usual care group (Active Comparator): We will provide patient education, home-based moderate to low-intensity rehabilitation
  Interventions: Behavioral: Disease and exercise suggestion
- CKD traditional rehabilitation group (Active Comparator): We will provide aerobic exercise, resistance exercise training, and patient education
  Interventions: Behavioral: Aerobic exercise; Behavioral: Resistance exercise; Behavioral: Disease and exercise suggestion
- CKD BFR group (Experimental): We will provide BFR combined with exercise and patient education
  Interventions: Behavioral: Aerobic exercise; Behavioral: Blood flow restriction; Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — The aerobic exercise intervention will utilize stationary bike. The program will be conducted 2 times per week over a 12 weeks
  Arms: CKD BFR group; CKD traditional rehabilitation group; healthy
Behavioral: Blood flow restriction — Blood flow restriction intervention will combined aerobic exercise and resistance exercise. The program will be conducted 2 times per week over a 12 weeks
  Arms: CKD BFR group; healthy
Behavioral: Resistance exercise — The resistance exercise will bilateral leg extension. The program will be conducted 2 times per week over a 12 weeks
  Arms: CKD BFR group; CKD traditional rehabilitation group; healthy
Behavioral: Disease and exercise suggestion — The participants will received self-care technique and home-based exercise approach
  Arms: CKD traditional rehabilitation group; CKD usual care group; healthy

SUMMARY:
Investigate the effects of exercise training on the cardiopulmonary function and exercise capacity in healthy and CKD patients

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a condition characterized by impaired kidney function lasting for more than 3 months, as estimated by the glomerular filtration rate (eGFR), which is classified into stages 1 to 5. Common symptoms include swelling, fatigue, and high blood pressure. Previous studies have indicated that physical inactivity in patients with CKD, often due to fatigue, leads to decreased physical fitness. In addition, secondary complications such as muscle mass loss and weakness are frequently observed, especially in the advanced stages of CKD.

To address this vicious cycle, aerobic and resistance training have been shown to mitigate these effects. Previous studies have reported that such exercise interventions can reduce fatigue and improve VO₂ peak in individuals with CKD. However, these exercise programs often involve high loads and frequencies, which may not be feasible for some CKD patients, particularly those with comorbidities such as diabetes or cardiovascular disease.

The effectiveness of blood flow restriction (BFR) exercise compared with high-load training has been demonstrated in older adults, showing improvements in functional ability and muscular adaptation. Therefore, the purpose of this study is to investigate the effects of incorporating blood flow restriction during exercise on cardiopulmonary function and exercise capacity in patients with CKD.

ELIGIBILITY:
Healthy

Inclusion Criteria:

• Aged 20~85 years old

Exclusion Criteria:

* Severe uncontrolled metabolic diseases (e.g., hyperthyroidism, diabetes, hypertension, hyperlipidemia, etc.)
* Severe pulmonary or cardiovascular diseases (e.g., pulmonary hypertension, chronic obstructive pulmonary disease (COPD), heart failure, cardiac arrhythmia)
* Presence of a cardiac pacemaker or a history of myocardial infarction within the past six months
* Severe musculoskeletal or neuromuscular disorders (e.g., advanced arthritis, limb amputation, post-polio syndrome, Parkinson's disease)
* Unstable vital signs (e.g., systolic blood pressure ≥180 mmHg, diastolic blood pressure ≥90 mmHg, requiring vasopressors, or resting heart rate >100 bpm)
* Prone to bruising
* Recent inflection < 1 month
* Pregnancy
* Kidney function impairment
* Cancer
* Simultaneously participating in other research

CKD

Inclusion criteria:

* Aged 20~85 years old
* eGFR< 90 ml/min/1.73 m2 over 3 months
* Stable condition without worsening in the past 3 months
* Ability to understand and follow verbal commends and cooperate with an exercise training program

Exclusion criteria:

* Severe uncontrolled metabolic diseases (e.g., hyperthyroidism, diabetes, hypertension, hyperlipidemia, etc.)
* Severe pulmonary or cardiovascular diseases (e.g., pulmonary hypertension, chronic obstructive pulmonary disease (COPD), heart failure, cardiac arrhythmia)
* Presence of a cardiac pacemaker or a history of myocardial infarction within the past six months
* Severe musculoskeletal or neuromuscular disorders (e.g., advanced arthritis, limb amputation, post-polio syndrome, Parkinson's disease)
* Unstable vital signs (e.g., systolic blood pressure ≥180 mmHg, diastolic blood pressure ≥90 mmHg, requiring vasopressors, or resting heart rate >100 bpm)
* Abnormal blood biochemical parameters (e.g., white blood cell count <2500/mm³, hemoglobin <8 mg/dL, total bilirubin >3 mg/dL, liver enzymes (GOT/AST, GPT/ALT) >3 times the upper limit of normal, platelet count <75,000/mm³
* Sensory or motor dysfunctions that affect walking ability
* Diagnosed systemic diseases under ongoing treatment (e.g., systemic lupus erythematosus, cancer, malignancies).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragm excursion and thickness | Change from baseline (0 week) to follow up (16 weeks)
  Diaphragm excursion (unit: mm) and thickness (unit: mm) are examined by diaphragmatic ultrasound when a participant performs maximal inspiration and expiration
Exercise capacity | Change form baseline (0 week) to follow up (16 weeks)
  A cardiopulmonary exercise test collects gases (including measures of oxygen consumption in ml/kg/min), which can be used to estimate exercise capacity

SECONDARY OUTCOMES:
Heart rate variability (Standard Deviation of Normal-to-Normal Intervals, SDNN) | Change form baseline (0 week) to follow up (16 weeks)
  Heart rate variability (HRV) is examined to assess the autonomic nervous system. Standard Deviation of Normal-to-Normal Intervals (SDNN, in ms)reflects overall heart rate variability and autonomic function
Heart rate variability (Root Mean Square of Successive Differences, RMSSD) | Change form baseline (0 week) to follow up (16 weeks)
  Root Mean Square of Successive Differences (RMSSD in ms) represents short-term HRV and parasympathetic activity
Heart rate variability (Low Frequency power, LF) | Change form baseline (0 week) to follow up (16 weeks)
  Low frequency power (LF, in ms²) reflects both sympathetic and parasympathetic modulation.
Heart rate variability (High Frequency power, HF) | Change from baseline (0 week) to follow-up (16 weeks)
  High frequency power (HF in ms²) reflects parasympathetic (vagal) activity.
Heart rate variability (LF/HF Ratio) | Change from baseline (0 week) to follow-up (16 weeks)
  LF/HF ratio represents sympathovagal balance.
Pulmonary function test | Change from baseline (0 week) to follow up (16 weeks)
  Pulmonary function test is examined by spirometry, which measures the ability to inhale and exhale air over time. The results include forced vital capacity (FVC in L), forced exploratory volume in the first second (FEV1 in L), and the FVC/FEV1 ratio.
Functional capacity | Change from baseline (0 week) to follow up (16 weeks)
  Functional capacity is examined by 6 minute walking test (6MWT, in m)
Functional ability | Change from baseline (0 week) to follow up (16 weeks)
  Functional ability is examined using the Timed Up and Go (TUG) test, where the time taken (in seconds) to complete the test is recorded.
Sit-and-Reach Test | Change from baseline (0 week) to follow up (16 weeks)
  Flexibility is examined by the sit and reach test (unit: cm).
Handgrip Strength | Change from baseline (0 week) to follow-up (16 weeks)
  Maximal voluntary handgrip strength. (unit: N)
Upper Limb Muscle Strength | Change from baseline (0 week) to follow up (16 weeks)
  Maximal voluntary contraction of upper limb muscles. (unit: N)
Neck Muscle Strength | Change from baseline (0 week) to follow up (16 weeks)
  Maximal voluntary contraction of neck muscles. (unit: N)
Knee Extensor Strength | Change from baseline (0 week) to follow-up (16 weeks)
  Maximal voluntary contraction of the knee extensor muscles. (unit: N)
Maximum respiratory pressure | Change from baseline (0 week) to follow up (20 weeks)
  Maximum respiratory pressure is measured using a manometer, which records both maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), in cmH₂O.
Fatigue Severity Scale (FSS) | Change form baseline (0 week) to follow up (16 weeks)
  the Fatigue Severity Scale (FSS) is a 7-point scale questionnaire that measures the patient's level of fatigue. It contains 9 questions, and a total score of 36 points or higher indicates that the patient may be experiencing clinically significant fatigue and requires further evaluation.
Kidney Disease Quality of Life (KDQOL) | Change form baseline (0 week) to follow up (16 weeks)
  The Kidney Disease Quality of Life (KDQOL) questionnaire is a standard tool for patients with kidney disease. It contains several subscales, and the raw scores are converted into normalized scores, with higher scores indicating better quality of life.
Modified Medical Research Council (mMRC) | Change from baseline (0 week) to follow up (16 weeks)
  The modified Medical Research Council (mMRC) dyspnea scale consists of 4 levels that describe respiratory difficulty during daily activities; higher levels indicate more severe symptoms.
Short Form-36 (SF-36) | Change from baseline (0 week) to follow up (16 weeks)
  The Short Form-36 (SF-36) measures physical and social health status, with higher scores representing better overall health

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ling Tasi, PhD, Principal Investigator — Department of Physical Therapy, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be decided after summarized data being published